CLINICAL TRIAL: NCT06205862
Title: Efficacy and Safety of Fecal Microbiota Transplantation in Reducing Recurrence of Colorectal Adenomas After Endoscopic Resection: a Multicenter, Open-label, Randomized Controlled Study
Brief Title: Efficacy and Safety of Fecal Microbiota Transplantation (FMT) in Reducing Recurrence of Colorectal Adenoma (CRA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Chen Ye, Professor, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20231219v2.6
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Fecal Microbiota Transplantation; Colorectal Adenoma; Gastrointestinal Microbiome
Keywords: Fecal Microbiota Transplantation; Colorectal Adenomas; Gastrointestinal Microbiome; Recurrence rate after endoscopic resection
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT group (Experimental): Participants are required to complete one colonoscopy and infuse 150ml of fecal suspension into the terminal ileum under endoscopy, performing the first fecal microbiota transplantation (FMT) on day 0. Subsequently, for 2 days continuously (day 1-2), the participants will undergo microbiota transplantation in the form of oral capsules, taking 40 FMT capsules within one day (20 capsules bid). Subsequently, participants will receive a maintenance treatment with oral FMT capsules (20 capsules bid) at 3, 6, and 9 months (approximately every 75 to 90 days). Participants will undergo their first follow-up colonoscopy between 6 to 12 months(the high-risk adenoma group will receive colonoscopy at 6 months, and the low-risk adenoma group will receive colonoscopy at 12 months).
  Interventions: Procedure: fecal microbiota transplantation
- No treatment group (No Intervention): Participants are required to complete one colonoscopy and during the procedure, 150ml of saline is infused into the terminal ileum on day 0. Subsequently, participants don't need any treatment. The participants will receive their first colonoscopy follow-up 6 to 12 months after enrollment.

INTERVENTIONS:
Procedure: fecal microbiota transplantation — We will use fecal suspensions and capsules prepared from the feces of healthy donors for fecal microbiota transplantation. Participants are required to complete one colonoscopy and infuse 150ml of fecal suspension into the terminal ileum under endoscopy, performing the first fecal microbiota transplantation (FMT) on day 0. Subsequently, for 2 days continuously (day 1-2), the participants will undergo microbiota transplantation in the form of oral capsules, taking 40 FMT capsules within one day (20 capsules bid). Subsequently, participants will receive a maintenance treatment with oral FMT capsules (20 capsules bid) at 3, 6, and 9 months (approximately every 75 to 90 days). Participants will undergo their first follow-up colonoscopy between 6 to 12 months(the high-risk adenoma group will receive colonoscopy at 6 months, and the low-risk adenoma group will receive colonoscopy at 12 months).
  Arms: FMT group

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of fecal microbiota transplantation in reducing recurrence of colorectal adenomas after endoscopic resection.

The main questions it aims to answer are:

* the efficacy and safety of fecal microbiota transplantation in reducing the recurrence rate of colorectal adenomas after endoscopic resection.
* changes in the intestinal and mucosal microbiota of patients before and after endoscopic treatment.
* changes in the intestinal and mucosal microbiota of patients before and after fecal microbiota transplantation.

Participants are required to complete one colonoscopy and infuse 150ml of fecal suspension into the terminal ileum under endoscopy, performing the first fecal microbiota transplantation (FMT) on day 0. Subsequently, for 2 days continuously (day 1-2), the participants will undergo microbiota transplantation in the form of oral capsules, taking 40 FMT capsules within one day (20 capsules bid). Subsequently, participants will receive a maintenance treatment with oral FMT capsules (20 capsules bid) at 3, 6, and 9 months (approximately every 75 to 90 days). Participants will undergo their first follow-up colonoscopy between 6 to 12 months(the high-risk adenoma group will receive colonoscopy at 6 months, and the low-risk adenoma group will receive colonoscopy at 12 months).

DETAILED DESCRIPTION:
Colorectal adenomas are precancerous lesions that can lead to colorectal cancer if not effectively managed. The standard treatment for colorectal adenomas is endoscopic resection. However, there is a significant rate of recurrence following this procedure, which poses a challenge for long-term management and prevention of colorectal cancer. Recent research has suggested a potential role for the gut microbiota in the development and recurrence of colorectal adenomas. Fecal microbiota transplantation (FMT) has been proposed as a novel strategy to manipulate the microbiota to reduce the recurrence of these lesions. This clinical trial aims to investigate both the efficacy and safety of FMT in reducing the recurrence of colorectal adenomas post endoscopic resection, and to elucidate the changes in intestinal and mucosal microbiota associated with the treatment.

The clinical trial is designed as a randomized controlled study where participants who have undergone endoscopic resection for colorectal adenomas are enrolled to receive FMT. The primary objective is to assess the efficacy of FMT in reducing the recurrence rate of colorectal adenomas. The secondary objective is to evaluate the safety of FMT in this patient population and to examine the changes in intestinal and mucosal microbiota before and after endoscopic treatment and FMT.

Participants are required to undergo a baseline colonoscopy to ensure the absence of residual adenomas post endoscopic resection. Following this, on day 0, participants will receive their first FMT via infusion of 150ml of fecal suspension into the terminal ileum under endoscopic guidance. This procedure aims to directly alter the gut microbiota by introducing a healthy donor's fecal material.

The FMT treatment is continued orally in the form of capsules for the next two days. Participants are instructed to ingest a considerable number of FMT capsules (40 capsules per day, 20 capsules twice daily) to maintain the introduced microbiota's presence and potential therapeutic effect.

After the initial intensive treatment phase, participants enter a maintenance phase where they receive oral FMT capsules at 3, 6, and 9 months (approximately every 75 to 90 days). This phase is designed to establish a newly balanced and potentially disease-modifying gut microbiome, allowing for a longitudinal assessment of the FMT's efficacy in reducing adenoma recurrence.

Safety assessments are performed throughout the trial, including monitoring for adverse events related to the FMT procedure and the overall health status of participants. Stool samples are collected at various time points to analyze changes in the gut microbiota composition using molecular techniques.

This clinical trial represents a critical step in understanding the potential role of FMT in preventing the recurrence of colorectal adenomas following endoscopic resection. By investigating both the efficacy and safety of FMT, as well as the associated changes in the gut microbiota, this study could significantly contribute to the development of novel therapeutic strategies for colorectal cancer prevention. If successful, this approach could provide a non-invasive and potentially effective treatment modality for patients at risk of recurrent colorectal adenomas, ultimately improving patient outcomes and reducing the burden of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, gender not specified.
2. Colorectal adenoma patients diagnosed by colonoscopy and treated with endoscopic resection (such as EMR, ESD, APC treatment, etc.)，or patients who have undergone endoscopic resection within the past 6 months and have pathologically confirmed colorectal adenoma.
3. Individuals who are able to swallow pills/capsules.
4. Individuals who voluntarily sign an informed consent form after fully understanding the purpose and procedures of this study, the characteristics of the disease, the therapeutic efficacy of the drugs, the related examination methods, and the potential risks/benefits of the study.

Exclusion Criteria:

1. Individuals in whom the adenoma was not completely removed in a previous colonoscopy;
2. Individuals who experienced serious complications during or after adenoma resection, including perforation, uncontrollable bleeding, or severe infection;
3. Individuals with a history of familial adenomatous polyposis (FAP) or hereditary nonpolyposis colorectal cancer (HNPCC/Lynch syndrome);
4. Individuals regularly taking aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase 2 (COX2) inhibitors, calcium, or vitamin D;
5. Individuals with a history of subtotal or total gastrectomy or partial bowel resection;
6. People who cannot tolerate colonoscopy;
7. Individuals with allergic diathesis, known allergies to fecal microbiota transplantation, drug allergies, or intolerance;
8. Individuals with serious heart, liver, or kidney diseases, or any history of cancer;
9. People suffering from severe constipation;
10. Pregnant women, breastfeeding mothers, or women planning to become pregnant;
11. Patients with mental illness who are unable to cooperate;
12. Individuals involved in the design, planning, or execution of this trial;
13. Any other individuals who, in the investigator's opinion, are unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
CRA recurrence rate | 6~12 months
  Percentage of patients who has recurrence of CRA(colorectal adenoma) during or after FMT.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0 | 1~12 months
  The number of participants with adverse events both severe and non-severe, assessed for severity based on the 5-grade criteria set by the NCI CTCAE version 5.0.
Intestinal Microbiota Composition Pre- and Post-FMT (Fecal Microbiota Transplantation) | 1~12 months
  Outcomes assessed included alpha and beta diversity, etc.
All polypoid lesions incidence rate | 6~12 months
  Percentage of patients who has incidence of all polypoid lesions during or after FMT.
CRC incidence rate | 6~12 months
  Percentage of patients who has incidence of CRC (colorectal cancer) during or after FMT.
Changes in intestinal mucosal microbiota Pre- and Post-FMT | 1~12 months
  Intestinal mucosal microbiota tests (16S rRNA gene sequencing, metagenome sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Ye Chen, MD, Principal Investigator — Shenzhen Hospital of Southern Medical University
Locations (5):
- China (5):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Luohu District People's Hospital, Shenzhen, Guangdong
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - Shunde Hospital of Southern Medical University, Shunde, Guangdong

IPD SHARING:
Plan to Share IPD: No